CLINICAL TRIAL: NCT04392648
Title: A Phase 1 Open-label Study to Evaluate the Safety, Tolerability and Efficacy of Intravenous TAK-573 as Part of Combination Therapy in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of Intravenous TAK-573 as Part of Combination Therapy in Participants With Relapsed or Refractory Multiple Myeloma (RRMM)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision (no enrollment)
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-573-1002; U1111-1249-1537 (Registry Identifier: WHO)
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: interventions — pomalidomide; Bortezomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Escalation:TAK-573 0.1-1.5mg/kg+Bortezomib+Dexamethasone (Experimental): TAK-573 0.1 to 1.5 milligram per kilogram (mg/kg), infusion, intravenously, once, every 3 weeks in a 21-days treatment cycle, along with bortezomib 1.3 milligram per square meter (mg/m^2), injection, subcutaneously, once on Days 1, 4, 8, and 11 and dexamethasone 40 milligram (mg) (20 mg if aged more than 75 years), tablets, orally on Days 1, 8, and 15 in each 21-days treatment cycle from Cycle 1 through Cycle 8. For participants who continue beyond Cycle 8, TAK-573 will be given as an infusion, intravenously, once, every 3 weeks in a 21-days treatment cycle with dexamethasone 40 mg (20 mg if aged more than 75 years), tablets, orally from Cycle 9 through Cycle 17.
  Interventions: Drug: TAK-573; Drug: Bortezomib; Drug: Dexamethasone
- Escalation:TAK-573 0.05-0.75mg/kg+Pomalidomide+Dexamethasone (Experimental): TAK-573 0.05 to 0.75 mg/kg, infusion, intravenously, once, every 4 weeks in a 28-days treatment cycle, along with pomalidomide 4 mg, capsules, orally, once daily from Days 1 through 21 and dexamethasone 40 mg (20 mg if aged more than 75 years), tablets, orally, once on Days 1, 8, 15, and 22 in each 28-days treatment cycle from Cycle 1 through Cycle 17.
  Interventions: Drug: TAK-573; Drug: Pomalidomide; Drug: Dexamethasone
- Escalation:TAK-573 0.1-1.5mg/kg+Cyclophosphamide+Dexamethasone (Experimental): TAK-573 0.1 to 1.5 mg/kg, infusion, intravenously, once, every 4 weeks in a 28-days treatment cycle, along with cyclophosphamide 300 mg/m^2, tablets, orally, once on Days 1, 8, and 15 and dexamethasone 40 mg (20 mg if aged more than 75 years), tablets, orally, once on Days 1, 8, 15, and 22 in each 28-days treatment cycle from Cycle 1 through Cycle 17.
  Interventions: Drug: TAK-573; Drug: Cyclophosphamide; Drug: Dexamethasone
- Expansion: TAK-573 + Bortezomib + Dexamethasone (Experimental): TAK-573, infusion, intravenously, once, every 3 weeks in a 21-days treatment cycle, along with bortezomib 1.3 mg/m^2, injection, subcutaneously, once on Days 1, 4, 8, and 11 and dexamethasone 40 mg (20 mg if aged more than 75 years), tablets, orally, once on Days 1, 8, and 15 in each 21-days treatment cycle until disease progression, intolerable toxicity, withdrawal from study, or death (up to 3 years). The dose of TAK-573 for Dose Expansion Phase will be the RP2D and recommended dose for expansion (RAD) determined in the previous Dose Escalation Phase.
  Interventions: Drug: TAK-573; Drug: Bortezomib; Drug: Dexamethasone
- Expansion: TAK-573 + Pomalidomide + Dexamethasone (Experimental): TAK-573, infusion, intravenously, once, every 4 weeks in a 28-days treatment cycle, along with pomalidomide 4 mg, capsules, orally, once daily from Days 1 through 21 and dexamethasone 40 mg (20 mg if aged more than 75 years), tablets, orally, once on Days 1, 8, 15, and 22 in each 28-days treatment cycle until disease progression, intolerable toxicity, withdrawal from study, or death (up to 3 years). The dose of TAK-573 for Dose Expansion Phase will be the RP2D and RAD determined in the previous Dose Escalation Phase.
  Interventions: Drug: TAK-573; Drug: Pomalidomide; Drug: Dexamethasone
- Expansion: TAK-573 + Cyclophosphamide + Dexamethasone (Experimental): TAK-573, infusion, intravenously, once, every 4 weeks in a 28-days treatment cycle, along with cyclophosphamide 300 mg/m^2, tablets, orally, once on Days 1, 8, and 15 and dexamethasone 40 mg (20 mg if aged more than 75 years), tablets, orally, once on Days 1, 8, 15, and 22 in each 28-days treatment cycle until disease progression, intolerable toxicity, withdrawal from study, or death (up to 3 years). The dose of TAK-573 for Dose Expansion Phase will be the RP2D and RAD determined in the previous Dose Escalation Phase.
  Interventions: Drug: TAK-573; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: TAK-573 — TAK-573 intravenous infusion.
Drug: Pomalidomide — Pomalidomide capsules orally.
  Arms: Escalation:TAK-573 0.05-0.75mg/kg+Pomalidomide+Dexamethasone; Expansion: TAK-573 + Pomalidomide + Dexamethasone
Drug: Bortezomib — Bortezomib injection subcutaneously.
  Arms: Escalation:TAK-573 0.1-1.5mg/kg+Bortezomib+Dexamethasone; Expansion: TAK-573 + Bortezomib + Dexamethasone
Drug: Cyclophosphamide — Cyclophosphamide tablets orally.
  Arms: Escalation:TAK-573 0.1-1.5mg/kg+Cyclophosphamide+Dexamethasone; Expansion: TAK-573 + Cyclophosphamide + Dexamethasone
Drug: Dexamethasone — Dexamethasone tablets orally.

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and recommended phase 2 dose (RP2D) of TAK-573 when used with dexamethasone and in combination with bortezomib, pomalidomide, or cyclophosphamide, in participants with RRMM.

DETAILED DESCRIPTION:
The drug that is being tested in this study is called TAK-573. The study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of TAK-573 when used in combination with dexamethasone and either bortezomib, pomalidomide or cyclophosphamide in participants with RRMM.

The study will be conducted in 2 phases: Dose Escalation Phase and Dose Expansion Phase. The study will enroll approximately 135 participants (approximately 60 participants in Dose Escalation Phase and approximately 75 participants in Dose Expansion Phase). The dose escalation phase will determine the recommended dose of TAK-573 along with the combination agents for the dose expansion phase.

This multi-center trial will be conducted in the United States, Germany, France, Spain, and Canada. The overall time to participate in this study is approximately 3 years. Participants will be followed up for 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Received >=2 prior lines of therapy, including treatment with lenalidomide and a proteasome inhibitor.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
3. With measurable disease, defined as at least 1 of the following:

   * Serum M protein >=500 mg/dL (>=5 gram per liter [g/L]) on serum protein electrophoresis (SPEP).
   * Urine M protein >=200 mg/24 hours on urine protein electrophoresis (UPEP).
   * Serum FLC assay result with an involved FLC level >=10 mg/dL (>=100 milligram per liter [mg/L]), provided the serum FLC ratio is abnormal.
4. Has adequate organ function as determined by the following laboratory values:

   * Absolute neutrophil count (ANC) >=1000 per cubic millimeter (/mm^3) (>=1.0*10^9 [per liter]/L)
   * Platelets >=75,000/mm^3 (>=75*10^9/L)
   * Hemoglobin >=80 g/L
   * Creatinine clearance >=30 milliliter per minute (mL/min)
   * Total serum bilirubin <=1.5*upper limit normal (ULN), >=2.0*ULN for participants with Gilbert's syndrome
   * Liver transaminases (alanine aminotransferase [ALT]/ aspartate aminotransferase [AST]) Serum ALT or AST <=3.0*ULN (<5*ULN if enzyme elevations are due to MM-related diffuse hepatic infiltrations).
5. Has received the final dose of any of the following treatments/procedures within the specified minimum intervals before first dose of TAK-573:

   * Chemotherapy, including proteasome inhibitors and immunomodulatory imide drug.(IMiDs) 14 days
   * Antimyeloma antibody therapy 21 days
   * Corticosteroid therapy for myeloma 7 days
   * Radiation therapy for localized bone lesions 7 days
   * Major surgery 21 days.

Exclusion Criteria:

1. Has polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin changes (POEMS) syndrome, monoclonal gammopathy of unknown significance, smoldering myeloma, solitary plasmacytoma, amyloidosis, Waldenström macroglobulinemia or IgM myeloma, lymphoplasmacytic lymphoma, or plasma cell leukemia.
2. Previous intolerance to combination agent.
3. For the pomalidomide expansion group only: no prior treatment with pomalidomide.
4. Inability to take prophylaxis needed for combination agent (deep vein thrombosis prophylaxis for pomalidomide, antiviral prophylaxis for proteasome inhibitor).
5. Who have received autologous stem cell transplant (SCT) within 60 days before first infusion of TAK-573 or participants who have received allogeneic SCT 6 months before first infusion. Graft-versus-host disease that is active or requires ongoing systemic immunosuppression.
6. Has not recovered from adverse reactions to prior myeloma treatment or procedures (chemotherapy, immunotherapy, radiation therapy) to NCI CTCAE Grade <=1 or baseline, except for sensory or motor neuropathy which should have recovered to Grade <=2 or baseline, Grade <2 for participants receiving bortezomib.
7. Has a chronic condition requiring the use of systemic corticosteroids >10 milligram per day (mg/day) of prednisone or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-24 (Estimated); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experienced at Least one Treatment Emergent Adverse Event (TEAE) | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
Number of Participants with Clinically Significant Vital Signs Values, Clinically Significant Change From Baseline in Clinical Laboratory Values and 12-lead Electrocardiograms (ECG), and who Received any Concomitant Medications | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
Dose Expansion Phase: Overall Response Rate (ORR) | Cycle 17 up to 3 years (Cycle length is equal to [=] 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  ORR is defined as the percentage of participants who achieved confirmed partial response (PR) or better during the study as assessed with International Myeloma Working Group (IMWG) Uniform Response Criteria. PR: greater than or equal to (>=) 50 percent (%) reduction of serum M protein and >=90% reduction in urine M-protein or less than (<) 200 milligram per 24 hour (mg/24 hour), or >=50% decrease in uninvolved free light chain (FLC). At baseline, a >=50% decrease in size of soft tissue plasmacytomas is required.

SECONDARY OUTCOMES:
Dose Escalation Phase, Cmax: Maximum Observed Serum Concentration for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, Tmax: Time to Reach the Maximum Serum Concentration (Cmax) for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, Lambda (λ) z: Apparent Serum Terminal Disposition Rate Constant for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, T1/2z: Apparent Serum Terminal Elimination Phase Half-life for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, CL: Total Clearance After Administration for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Dose Escalation Phase, Vss: Volume of Distribution at Steady State After Administration for TAK-573 | Cycles 1 and 2 Day 1: pre-dose and at multiple time points (up to 336 hours) post-dose (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
Percentage of Participants with Positive Antidrug Antibodies (ADA) for Anti-573 | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length is = 21 days in Arm 4 and = 28 days in Arms 5 and 6)
Dose Escalation Phase: ORR | Up to Cycle 17 (Cycle length = 21 days in Dose Escalation Phase Arm 1 and is = 28 days in Dose Escalation Phase Arms 2 and 3)
  ORR is defined as the percentage of participants who achieved confirmed PR or better during the study as assessed with IMWG Uniform Response Criteria. PR: >= 50% reduction of serum M protein and >=90% reduction in urine M-protein or <200 mg/24 hour, or >=50% decrease in uninvolved FLC. At baseline, a >=50% decrease in size of soft tissue plasmacytomas is required.
Best Overall Response (BOR) | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  BOR is defined as the best response recorded after the first dose of any study drug until subsequent therapy for multiple myeloma (MM). BOR will be assessed as per IMWG uniform response criteria.
Clinical Benefit Rate (CBR) | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  The CBR is defined as the percentage of participants who achieved an ORR along with the minimal response (MR) or better during the study as assessed with IMWG Uniform Response Criteria. ORR is defined as the percentage of participants who achieved confirmed PR or better during the study as assessed with IMWG Uniform Response Criteria. MR is defined as a >=25% but less than or equal to (<=) 49% reduction of serum M protein and reduction in 24-hour urine M protein by 50% to 89%. In addition, if present at baseline, 25% to 49% reduction in size of soft tissue plasmacytomas is also required. No increase in size or number of lytic bone lesions (development of compression fracture does not exclude response).
Disease Control Rate (DCR) | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  The DCR is defined as the percentage of participants who achieved CBR along with a stable disease (SD) or better during the study as assessed with IMWG Uniform Response Criteria. The CBR is defined as the percentage of participants who achieved an ORR along with the minimal response (MR) or better during the study as assessed with IMWG Uniform Response Criteria. SD is defined as no known evidence of progressive or new bone lesions.
Median Duration of Response (DOR) | Dose Escalation Phase: up to Cycle 17 (Cycle length = 21 days in Arm 1 and is = 28 days in Arms 2 and 3); Dose Expansion Phase: Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  DOR: number of days from first documentation of a confirmed response until progressive disease (PD) or until last adequate response assessment if there is no PD. DOR will be assessed as per IMWG uniform response criteria. PD: increase of 25% from lowest response value in any one or more of the following: serum M protein and/or; urine M component and/or; only in participants without measurable serum and urine M protein levels; the difference between involved and uninvolved FLC levels (absolute increase >10 milligram per deciliter [mg/dL]); Bone marrow plasma cell percentage (absolute percentage must be >10%); definite development of new bone lesions or soft tissue plasmacytomas or increase in the size of existing bone lesions/soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Dose Expansion Phase: Progression Free Survival (PFS) | Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  PFS: time from date of first dose until sooner of the date of PD, defined by IMWG criteria, or the date of death due to any cause, whichever occurs first. PD: increase of 25% from lowest response value in any one or more of the following: serum M protein and/or; urine M component and/or; only in participants without measurable serum and urine M protein levels; the difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL); Bone marrow plasma cell percentage (absolute percentage must be >10%); definite development of new bone lesions or soft tissue plasmacytomas or increase in the size of existing bone lesions/soft tissue plasmacytomas; development of hypercalcemia that can be attributed solely to plasma cell proliferative disorder.
Dose Expansion Phase: Time to Response (TTR) | Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  TTR is defined as the time from first dose to the date of first documentation of response (PR or better). PR: A >=50% reduction of serum M protein and >=90% reduction in urine M-protein or <200 mg/24 hour, or >=50% decrease in uninvolved FLC. A >=50% decrease in size of soft tissue plasmacytomas present at baseline. The Kaplan-Meier method will be used to estimate the distribution of TTR for dose level and group with at least 10 participants in the safety analysis set.
Dose Expansion Phase: Overall Survival (OS) | Cycle 17 up to 3 years (Cycle length = 21 days in Arm 4 and is = 28 days in Arms 5 and 6)
  OS is defined as the time elapsed between the date of diagnosis until death, with censoring of participants who are alive when last seen or who are lost to follow up.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit USMedInfo@tevapharm.com to make your request.